CLINICAL TRIAL: NCT07333261
Title: A Phase 1b Study of BMS-986453, Dual Targeting BCMAxGPRC5D Chimeric Antigen Receptor T Cells, in Participants With Newly Diagnosed Multiple Myeloma
Brief Title: Study of BMS-986453 in Newly Diagnosed Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Susan Bal (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Susan Bal, Associate Professor, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300015643 (UAB2595); 000551303 (Other: BMS)
Record Dates: First submitted 2025-12-02; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: This is a single center, open-label, Phase 1b study to determine the safety, and preliminary efficacy of BMS-986453, a dual targeting CAR-T cell product targeting BCMA and GPRC5D, in participants with NDMM in whom ASCT is not planned.
  The study will evaluate the safety, PK, pharmacodynamic, and preliminary efficacy of BMS-986453 at the RP2D. All treated participants will complete three periods: pre-treatment, treatment, and post- treatment follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose BMS-986453 (Experimental): Participants will be treated with fludarabine IV (30 mg/m2/day) and cyclophosphamide IV (300 mg/m2/day) for 3 days prior to BMS-986453 infusion.
  A single dose of BMS-986453 administered by IV infusion.
  Interventions: Drug: BMS-986453

INTERVENTIONS:
Drug: BMS-986453 — Will be given as a single dose administered by IV infusion.

SUMMARY:
This is a phase 1b study evaluating if BMS-986453 is safe and effective in treating people who have newly diagnosed multiple myeloma after completing initial therapy (induction) when a stem cell transplant is not intended.

DETAILED DESCRIPTION:
This is an open-label study. The investigators propose to examine if BMS-986453 in people with newly diagnosed multiple myeloma may help control their disease for a prolonged period of time despite one-time treatment and challenge continuous treatment which is otherwise prescribed.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years with no upper age limit
2. NDMM with indication for initiation of therapy diagnosed within last 12 months. Pretreatment parameters necessary for disease characterization and response assessment must be available.
3. Not eligible for ASCT by institutional criteria or deferring ASCT due to personal preference.
4. ECOG performance status 0-1
5. Adequate organ function

Exclusion Criteria:

1. Known active or history of central nervous system (CNS) involvement of MM.
2. Plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS or clinically significant amiloidosis.
3. Prior history of other malignancies
4. Uncontrolled infection

Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2043-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Baseline up to 5 years
  Evaluate the safety and tolerability of BMS-986453 in participants with NDMM.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Baseline up to 5 years
  Measure of clinical response.
Overall Survival (OS) | Baseline up to 5 years
  Measure of clinical response.
Progression Free Survival (PFS) | Baseline up to 5 years
  Measure of clinical response.
Pharmacokinetics (PK) | Baseline up to 2 years
  Measures of observed blood concentration of BMS-968453.
Complete response rate | Baseline up to 5 years
  Measures of clinical response.
MRD negativity | Baseline up to 5 years
  Proportion of participants with overall MRD negativity, 9-month MRD negativity rates as well as sustained (>12 months) MRD negativity.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 15 years
  Assess long-term toxicity
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 15 years
  Assess lentiviral vector safety
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 15 years
  Assess disease status
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 15 years
  Assess survival after BMS-968453 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bal, MD, Principal Investigator — The University of Alabama at Birmingham; Luciano A Costa, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States